CLINICAL TRIAL: NCT05582161
Title: Efficacy Biomarkers of DAOIB for Dementia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202101070A3
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAOIB (Experimental)
  Interventions: Drug: DAOIB

INTERVENTIONS:
Drug: DAOIB — The DAOIB dose will be adjusted every 8 weeks according to clinical evaluation.

SUMMARY:
This open-label clinical trial will enroll patients with aMCI or mild AD, and they will be treated with DAOIB for 24 weeks. We will assess the patients before entering the study, 8 weeks, 16 weeks, and end point (24 weeks) of the study, and measure blood NMDA and oxidative stress - related biomarkers every 8 weeks. We hypothesize that NMDA and oxidative stress - related biomarkers can predict the efficacy of DAOIB for patients with aMCI or mild AD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's disease or mild cognitive impairment
* MMSE between 10-26
* CDR 1 or 0.5

Exclusion Criteria:

* Hachinski Ischemic Score > 4
* Substance abuse/dependence
* Parkinson disease, epilepsy, dementia with psychotic features
* Major depressive disorder
* Major physical illnesses
* Severe visual or hearing impairment

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's disease assessment scale - cognitive subscale at week 8, 16 and 24 | week 0, 8, 16, 24
  Alzheimer's disease assessment scale-cognitive subscale scores range from 0 (best) to 70 (worst)

SECONDARY OUTCOMES:
Change from baseline in the composite score of a battery of additional cognitive tests at week 24 | week 0, 24
  The battery of additional cognitive tests include speed of processing (Category Fluency), working memory (Wechsler Memory Scale, Spatial Span), verbal/nonverbal learning and memory tests (Wechsler Memory Scale, Word Listing)
Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24 | week 8, 16, 24
  Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24
Change from baseline in Alzheimer's disease Cooperative Study scale for ADL in MCI (ADCS-MCI-ADL) score at week 8, 16 and 24 | week 0, 8, 16, 24
  The assessment appears to be a suitable instrument for evaluating activities of daily living in early-phase dementia. Its scores range from 0 (worst) to 78 (best)
Change from baseline of Geriatric Depression Scale | week 0, 8, 16, 24
  Assessment of geriatric depressive symptoms
Change from baseline in Mini-Mental Status examination score at week 8, 16 and 24 | week 0, 8, 16, 24
  Change from baseline in Mini-Mental Status examination score at week 8, 16 and 24

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No